CLINICAL TRIAL: NCT06418087
Title: A Multicenter Phase II, Single Arm Study of Durvalumab (MEDI 4736) With Carboplatin Plus Etoposide for 4 Cycles Followed by Durvalumab Maintenance in Patients With Metastatic Pulmonary Large-cell Neuroendocrine Carcinoma (LCNEC)
Brief Title: Durvalumab With Carboplatin and Etoposide Chemotherapy in Pulmonary Large-cell Neuroendocrine Carcinoma (LCNEC)
Acronym: DUPLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUPLE- GOIRC- 05-2020
Record Dates: First submitted 2022-08-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Large-cell Neuroendocrine Carcinoma
MeSH Terms: interventions — durvalumab; Solutions; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Pulmonary Large-cell Neuroendocrine Carcinoma (Experimental): All enrolled patients will receive intravenous infusion of durvalumab 1500 mg on day 1 (induction phase) with carboplatin (AUC 5 on day 1), etoposide (100 mg/sqm on days 1-3) every 3 weeks, and durvalumab (1500 mg on day 1) administered every three weeks for up to 4 cycles (induction phase) or until progression of disease, unacceptable toxicity, patient refusal or loss of clinical benefit (for durvalumab). Treatment with intravenous durvalumab (1500 mg on day 1) every 4 weeks ± 3 days (maintenance phase) will continue until completion of 24 courses (for a total of 28 courses, including the 4 courses of induction phase) or 2 years of treatment whichever occurs first, disease progression, unacceptable toxicity, patient refusal or loss of clinical benefit.
  Interventions: Drug: Durvalumab 50 MG/1 ML Intravenous Solution [IMFINZI]

INTERVENTIONS:
Drug: Durvalumab 50 MG/1 ML Intravenous Solution [IMFINZI] — Intravenous infusion of durvalumab 1500 mg on day 1 (induction phase) with carboplatin (AUC 5 on day 1), etoposide (100 mg/sqm on days 1-3) every 3 weeks, and durvalumab (1500 mg on day 1) administered every three weeks for up to 4 cycles (induction phase) or until progression of disease, unacceptable toxicity, patient refusal or loss of clinical benefit (for durvalumab).
  Treatment with intravenous durvalumab (1500 mg on day 1) every 4 weeks ± 3 days (maintenance phase) will continue until completion of 24 courses (for a total of 28 courses, including the 4 courses of induction phase) or 2 years of treatment whichever occurs first, disease progression, unacceptable toxicity, patient refusal or loss of clinical benefit.
  Other Names: Carboplatino AHCL 10 mg/ml Concentrate for solution for infusion; Etoposide 20 mg/ml Concentrate for solution for infusion

SUMMARY:
A prospective multicenter, single-arm phase II study enrolling treatment-naïve patients with metastatic pulmonary large-cell neuroendocrine carcinoma (LCNEC)

DETAILED DESCRIPTION:
This is a prospective multicenter, single-arm phase II study enrolling treatment-naïve patients with metastatic pulmonary large-cell neuroendocrine carcinoma (LCNEC). Enrolled subjects will receive a combination of intravenous carboplatin (AUC 5 on day 1), etoposide (100 mg/sqm on days 1-3), and durvalumab (1500 mg on day 1) administered every three weeks for a total of 4 courses (induction phase) or until progression of disease, unacceptable toxicity, patient refusal or loss of clinical benefit. Treatment with intravenous durvalumab (1500 mg on day 1) every 4 weeks (maintenance phase) will continue until completion of 24 courses (for a total of 28 courses, including the 4 courses of induction phase) or 2 years of treatment whichever occurs first, disease progression, unacceptable toxicity, patient refusal or loss of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Age ≥18 years at the time of study entry
* Histologically or cytologically (cell blocks only; smears are not acceptable) documented pulmonary large-cell neuroendocrine carcinoma (LCNEC)
* Stage IV disease or unresectable stage IIIB, which cannot be safely encompassed in a single RT field (e.g. supraclavicular N3, T4 by infiltration of vertebral body), according to the AJCC 8th edition Cancer Staging Manual
* Body weight >30 kg
* No prior chemotherapy or treatment with another systemic anti-cancer agent. Patients who have received prior chemoradiotherapy for locally advanced pulmonary LCNEC must have been treated with curative intent and experienced a treatment-free interval of at least 6 months from last chemotherapy, radiotherapy or chemoradiotherapy cycle to disease relapse, progression, or diagnosis of metastatic LCNEC. In this case, all toxicity from previous treatments should be resolved and no cumulative toxicity of grade >1 should be present (see also Section 4.2 "Exclusion criteria").
* No need for concomitant chest irradiation
* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* At least one lesion measurable according to RECIST v 1.1 outside of the CNS, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements
* Adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1500/µL, hemoglobin ≥9 g/dL (5.58 mmol/L), and platelets ≥100,000/µL.
* Adequate hepatic and renal functions:
* Total bilirubin < 1.5 times the upper limits of normal [ULN]
* AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
* Serum creatinine ≤1.5 times the ULN or creatinine clearance, calculated according to the formula of Cockcroft and Gault > 60 ml/min
* The patient has adequate coagulation function as defined by International Normalized Ratio (INR) ≤1.5 and a partial thromboplastin time (PTT) (PTT/aPTT) < 1.5 x ULN.). Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). If receiving warfarin, the patient must have an INR ≤3.0.
* Female patients must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
* Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
* Women under 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 6 months after the last dose of chemotherapy or 90 days after the last dose of durvalumab, whichever occurs last. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, and vasectomized partner (on the understanding that this is the only one partner during the whole study duration).
* Male patients who are sexually active must be willing to use barrier contraceptives (i.e., by use of condoms) during sex with all partners during treatment with chemotherapy and for at least 6 months after the final dose of chemotherapy or 90 days after the last dose of durvalumab, whichever occurs last, to avoid exposing the embryo. Men must refrain from donating sperm during this same period
* Ability to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

* Symptomatic brain metastases or spinal cord compression (CT or MRI of the head is required within 4 weeks prior to randomization) requiring immediate radiotherapy for palliation. Patients with asymptomatic CNS lesions are eligible, provided that all of the following criteria are met:
* The patient has no history of intracranial hemorrhage, spinal cord hemorrhage or hemorrhagic intracranial lesions
* At least 14 days between the end of stereotactic radiotherapy or whole brain radiotherapy and initiation of study treatment, or at least 28 days between neurosurgical resection and initiation of study treatment
* The patient is on a dose of corticosteroids ≤ 10 mg of oral prednisone or equivalent; anticonvulsant therapy at a stable dose is permitted
* Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla or spinal cord)
* There is no evidence of interim progression between completion of CNS directed therapy (if administered) and initiation of study treatment
* History of leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Patients with indwelling catheters (e.g., Pleura-Cath) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected calcium > ULN)
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C
* Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
* Patients positive for hepatitis C (HCV) antibody are eligible if polymerase chain reaction is negative for HCV RNA.
* Significant traumatic injury or radiotherapy involving an extensive field within the last 4 weeks prior to first dose of study treatment or anticipation of the need for major surgery during study treatment. Palliative radiotherapy to a limited field is allowed if concluded at least 2 weeks prior enrolment.
* Other malignancies (previous or current), except for adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, localized prostate cancer surgically treated with curative intent or ductal carcinoma in situ treated surgically treated with curative intent or if previous malignancy was more than 5 years prior and there are no signs or symptoms of recurrence
* Major surgery (including open biopsy) within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to the first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
* Prior allogeneic stem cell or solid organ transplantation.
* Patients with any underlying medical condition that might be aggravated by treatment or which cannot be controlled i.e. patients with active serious infection, uncontrolled diabetes mellitus, pericardial effusion.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment other than those in the present study. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Treatment with any other investigational agent within 30 days prior to starting study treatment, or concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Patients with celiac disease controlled by diet alone
* History or active autoimmune neurologic paraneoplastic syndrome (e.g. non-infectious encephalitis, Lambert-Eaton syndrome etc.) or any other immune-mediated paraneoplastic syndrome.
* Patients with SIADH or ectopic ATCH production are allowed on trial
* Patient has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* History of idiopathic pulmonary fibrosis, including pneumonitis, drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Prior therapy with any anti-PD-1, anti-PD-L1including durvalumab, or anti-PD-L2 agent and anti-CTL-A4 agent.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment.
* Any condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of randomization. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* History of allergies or hypersensitivity to any study drugs or study drug components or CHO derived products.
* The patient is pregnant or breast-feeding
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with carboplatin, etoposide or durvalumab may be included only after consultation with the Study Physician.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 6 months after last chemotherapy dose or 90 days after the last dose of durvalumab, whichever occurs last. Patients should refrain from donating sperm from the start of dosing until 4 months after discontinuing study treatment.
* Patients should not donate blood whilst on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the combination of carboplatin + etoposide + durvalumab in treatment-naïve patients, as first line treatment, with metastatic pulmonary LCNEC | 1 year
  Efficacy of the combination of carboplatin + etoposide Overall Survival rate at 1 year

SECONDARY OUTCOMES:
Activity of the combination of carboplatin + etoposide + durvalumab as first-line treatment for patients with metastatic pulmonary LCNEC | 1 year
  Activity of the combination of carboplatin + etoposide + durvalumab as first-line treatment for patients with metastatic pulmonary LCNEC Median OS PFS ORR DCR and DoR at 1 year
Number of Participants with treatment-related Adverse Events as assessed by CTCAE v. 5.0 - The safety and tolerability profile of the combination of carboplatin + etoposide + durvalumab as first-line treatment for patients with metastatic pulmonary LCNEC | 1 year
  Safety and tolerability profile of the combination of carboplatin + etoposide + durvalumab as first-line treatment for patients with metastatic pulmonary LCNEC

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, Study Director — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (15):
- Italy (15):
  - IRCCS AOU Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Istituto Oncologico del Mediterraneo IOM - Viagrande Catania, Viagrande, CT
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l. IRCCS, Meldola, FC
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Humanitas Research Hospital, Rozzano, MI
  - Istituto Oncologico Veneto IRCCS-IOV, Padua, PD
  - Centro di riferimento oncologico di Aviano, Aviano, PN
  - Azienda Ospedaliera San Camillo Forlanini-Ospedale San Camillo, Roma, RM
  - AOU Sassari - Ospedale SS. Annunziata, Sassari, SS
  - AOU Ospedale San Luigi Gonzaga, Orbassano, TO
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico Bari, Bari
  - Azienda Usl Toscana nord ovest Ospedale San Luca, Lucca
  - Ospedale San Gerardo Monza, Monza
  - A.O.R.N. "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria di Parma, Parma